CLINICAL TRIAL: NCT02361801
Title: Liberal Versus Restrictive Dobutamine in Cardiac Surgery (DOBUTACS): a Prospective Randomized Non-inferiority Clinical Trial
Brief Title: Liberal Versus Restrictive Use of Dobutamine in Cardiac Surgery
Acronym: DOBUTACS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ludhmila Abrahão Hajjar MD, PhD, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DOBUTACS
Record Dates: First submitted 2015-02-02; First posted 2015-02-12 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Cardiac Output, Low; Coronary Disease
Keywords: cardiac surgery; dobutamine
MeSH Terms: conditions — Cardiac Output, Low; Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal dobutamine group (Active Comparator): All patients will receive dobutamine at the cardiopulmonary bypass weaning
  Interventions: Drug: Liberal dobutamine protocol
- Restrictive dobutamine group (Active Comparator): Patients will only receive dobutamine if they present clinical signs of cardiogenic shock
  Interventions: Drug: Restrictive dobutamine protocol

INTERVENTIONS:
Drug: Liberal dobutamine protocol — All patients will receive dobutamine at the cardiopulmonary bypass weaning.
  Arms: Liberal dobutamine group
Drug: Restrictive dobutamine protocol — Patients will receive dobutamine during the first 8 hours after cardiopulmonary bypass weaning only if they have a cardiac index of ≤ 2.5L/min/m2 and at least one sign of tissue hypoperfusion: ScvO2 ≤ 70% and / or urine output < 2 mL/Kg/h despite adequate fluid replacement.
  Arms: Restrictive dobutamine group

SUMMARY:
Inotropic agents are usually administered in the postoperative period after cardiac surgery. In most cases, dobutamine is administered routinely, for the probable occurrence of myocardial dysfunction after cardiopulmonary bypass or a low cardiac output with minimal evidence of altered tissue perfusion.

Recent data show that inotropic agents are used in 35-52% of cardiac surgeries in the perioperative period. However, the use of inotropic agents may be associated with adverse events, including myocardial ischemia, by elevation in myocardial oxygen consumption and the imbalance between supply and consumption, and tachyarrhythmias (atrial fibrillation, sinus tachycardia, ventricular tachyarrhythmias), primarily due to the β1-adrenergic effect.

This study is a non-inferiority clinical randomized study aiming to compare the use of dobutamine in a liberal strategy (in all patients at the time of withdrawal of CPB) with a restrictive strategy (based on clinical and hemodynamic evidence of low cardiac output syndrome associated with altered tissue perfusion). Our primary hypothesis is that the restrictive use of dobutamine is as safe and effective as the liberal one.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery of coronary artery bypass graft (CABG) with cardiopulmonary bypass;
* Age equal or greater than 18 years;
* Written informed consent.

Exclusion Criteria:

* Previous ventricular dysfunction (ejection fraction lower than 50%)
* Sustained supraventricular or ventricular arrhythmias;
* Cardiogenic shock or need for inotropes before surgery;
* Immediate need of ventricular assist device or intraaortic balloon after CPB;
* Combined procedure;
* Pregnancy;
* Participation in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Combined endpoint of arrhythmias (ventricular and supraventricular), acute myocardial infarction, stroke or transient ischemic attack, low-output syndrome, cardiogenic shock and death from all causes within 30 days after cardiac surgery | 30 days

SECONDARY OUTCOMES:
Mortality rate | 30 days
  We will compare the mortality rate between groups within 30 days after randomization
Acute myocardial infarction incidence | 30 days
  We will compare the incidence of acute myocardial infarction between groups within 30 days after randomization
Stroke incidence | 30 days
  We will compare the incidence of stroke between groups within 30 days after randomization
Low cardiac output syndrome | 30 days
  We will compare the incidence of low cardiac output syndrome between groups within 30 days after randomization
Cardiogenic shock | 30 days
  We will compare the incidence of cardiogenic shock between groups within 30 days after randomization
Cardiac arrhythmias | 30 days
  We will compare the incidence of ventricular and supraventricular arrhythmias between groups within 30 days after randomization
ICU and hospital length of stay | 30 days
Days free of mechanical ventilation | 30 days
  We will compare the number of days free of mechanical ventilation between groups within 30 days after randomization
Severe sepsis and septic shock | 30 days
  We will compare the incidence of severe sepsis and septic shock between groups within 30 days after randomization
SOFA score within 72 hours | 72 hours
  We will compare the SOFA score between groups 72 hours after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Franco RA, de Almeida JP, Landoni G, Scheeren TWL, Galas FRBG, Fukushima JT, Zefferino S, Nardelli P, de Albuquerque Piccioni M, Arita ECTC, Park CHL, Cunha LCC, de Oliveira GQ, Costa IBSDS, Kalil Filho R, Jatene FB, Hajjar LA. Dobutamine-sparing versus dobutamine-to-all strategy in cardiac surgery: a randomized noninferiority trial. Ann Intensive Care. 2021 Jan 26;11(1):15. doi: 10.1186/s13613-021-00808-6. PMID 33496877